CLINICAL TRIAL: NCT03081494
Title: Phase Ib Study of PDR001 in Combination With Regorafenib in Adult Patients With Previously Treated Metastatic Microsatellite Stable (MSS) Colorectal Cancer
Brief Title: Phase Ib Study of PDR001 in Combination With Regorafenib in Adult Patients With Previously Treated Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CPDR001I2102; 2017-000466-30 (EudraCT Number)
Record Dates: First submitted 2017-03-10; First posted 2017-03-16 (Actual); Last update posted 2020-12-11 (Actual); Status verified 2020-12

CONDITIONS: Metastatic Colorectal Cancer
Keywords: PDR001; MCC; immunotherapy; regorafenib; CRC; MMS; CMS4; ElevatION:CRC-102
MeSH Terms: conditions — Colorectal Neoplasms | interventions — spartalizumab; regorafenib

STUDY DESIGN:
Intervention Model Description: Phase 1b study, dose escalation (N=~12). One single arm: PDR001 in combination with regorafenib
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- spartalizumab (PDR001) + regorafenib (Experimental): Subjects with metastatic MSS CRC received a combination of spartalizumab and regorafenib.
  Interventions: Drug: spartalizumab (PDR001); Drug: regorafenib

INTERVENTIONS:
Drug: spartalizumab (PDR001) — 100 mg lyophilisate in vial received 400 mg every 4 weeks
  Other Names: PDR001
Drug: regorafenib — 120 mg once daily first 21 days of each 28-day cycle (=4 weeks)

SUMMARY:
This was a phase Ib study of PDR001 in combination with regorafenib in adult patients with previously treated metastatic microsatellite stable (MSS) colorectal cancer. The study assessed primarily the safety and tolerability of PDR001 in combination with regorafenib.

ELIGIBILITY:
Key inclusion criteria:

1. Patients with metastatic colorectal adenocarcinoma.
2. Patients must provide a newly obtained or an archival tumor sample corresponding to CRC diagnosis (primary tumor) with sufficient tissue quality (qualified) for analysis
3. Patients must provide a newly obtained tumor tissue sample from a metastatic site
4. Patients with the presence of at least one lesion with measurable disease as per RECIST
5. Patients previously treated with two prior regimen as per standard of care and have experienced disease progression (including -VEGF and EGFR targeted therapies (if KRAS wild).
6. Patient has an Eastern Cooperative Oncology Group (ECOG) performance status 0-1

Key exclusion criteria:

1. Patients with MSI-H colorectal adenocarcinoma as defined per local assessment using standard of care testing
2. Patients with metastatic disease amenable to be resected with potentially curative surgery
3. Patients who have had chemotherapy, radiation, or biological cancer therapy within 14 days prior to the first dose of study treatment
4. Patients with a history of prior treatment with anti-PD-1, anti-PD-L1, anti-PDL2, anti- CTLA-4 antibodies, other checkpoint inhibitors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-06-09 (Actual); Primary Completion 2019-05-07 (Actual); Study Completion 2019-05-07 (Actual)

PRIMARY OUTCOMES:
Incidence of Dose-limiting toxicity (DLT) | 8 Weeks
  A dose-limiting toxicity (DLT) was defined as (1) an adverse event or abnormal laboratory value (assessed as unrelated to disease, disease progression, inter-current illness, or concomitant medications) that occurred within the first 8 weeks (56 days) of treatment with PDR001 in combination with regorafenib during dose escalation part and (2) met any of the pre-defined criteria.

SECONDARY OUTCOMES:
Incidence of adverse events (AEs) and serious adverse events (SAEs) | Up to 150 days after last administration of PDR001
  Incidence of all treatment-emergent adverse events (including clinically significant changes in laboratory values, vital signs and ECG), as assessed by CTCAE v4.03.
Severity of AEs and SAEs | Up to 150 days after last administration of PDR001
  Severity including dose interruptions and reductions.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (11):
- Australia (2):
  - Novartis Investigative Site, St Leonards, New South Wales
  - Novartis Investigative Site, Murdoch, Western Australia
- Novartis Investigative Site, Montreal, Quebec, Canada
- Novartis Investigative Site, Tel Aviv, Israel
- Italy (2):
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Rozzano, MI
- Novartis Investigative Site, Leiden, Netherlands
- Novartis Investigative Site, Singapore, Singapore
- Novartis Investigative Site, Seoul, Korea, South Korea
- Spain (2):
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Madrid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Novartis results database — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=17553
- See also: A Plain Language Trial Summary is available on novartisclinicatrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=553